CLINICAL TRIAL: NCT04560764
Title: Virtual Reality and Action-Observation Therapy: An Integrated Approach Supported by Novel Technologies for Upper Limb Impairment in Subacute Stroke
Brief Title: Physiotherapy and Action-Observation Therapy: An Integrated Approach for Upper Limb Impairment in Subacute Stroke
Acronym: PHOENICS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes in the rehabilitation service that no longer allowed the recruitment of patients
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Riccardo Buraschi, Principal investigator, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDG_AOTVR
Record Dates: First submitted 2019-10-02; First posted 2020-09-23 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Stroke
Keywords: Upper limb impairment; Virtual Reality; Action Observation Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality + Action Observation Therapy (Experimental): Participants will see a video demonstrating the exercise they will be later asked to perform. The same procedure is performed for each of the four different exercises.
  Interventions: Device: Virtual Reality; Device: Action Observation Therapy; Other: Standard treatment
- Virtual Reality + Landscape video (Sham Comparator): Participants will see a video demonstrating a natural landscape and later they will perform an exercise. The same procedure is performed for each of the four different exercises.
  Interventions: Device: Virtual Reality; Device: Landscape video; Other: Standard treatment

INTERVENTIONS:
Device: Virtual Reality — Participants in both groups will attend 10 sessions of approximately 30 minutes each three times a week. Each session contemplates the execution of a single repetition of two minutes of each of the four exercises.
  There are four exercises:
  1. Reaching: the participant is requested to reach a target in front of him with the paretic hand; the target will appear in a different place every time;
  2. Reaching and grasping: the participant is requested to grab a wooden cube with the paretic hand and place it into a bowl positioned in front of him; the cube will appear in a different place every time;
  3. Goalkeeper: the participant is requested to block a ball coming towards him with the paretic hand; the ball will appear in a different place every time;
  4. Occupational task: the participant is requested to grab four cans, one at time, with the paretic hand and place them on four targets placed on a hemispherical arch.
  Each exercise provides six levels of increasing difficulty.
Device: Action Observation Therapy — Before the execution of the exercises described in the intervention "Virtual Reality", the participants in the experimental group will see a video demonstrating the same exercise (according to the level of difficulty selected) he will be later asked to perform for two minutes.
  Arms: Virtual Reality + Action Observation Therapy
Device: Landscape video — Before the execution of the exercises described in the intervention "Virtual Reality", the participants in the sham comparator group will see a video of a natural landscape for two minutes.
  Arms: Virtual Reality + Landscape video
Other: Standard treatment — Participants in both groups will receive the standard treatment, one hour a day for three days a week.

SUMMARY:
Motor impairment is one of the most common result of a stroke, which causes disability and difficulties in activities of daily living. This motor impairment can concern the upper limb or the lower limb, or both. Several studies investigates the efficacy of different treatment approaches on upper limb and hand function. None of them combined exercise in a virtual context with Action Observation Therapy, consisting in watching an action before doing it.

This study evaluates the addition of Action Observation Therapy (AOT) to Virtual Reality (VR) in the rehabilitation of upper limb impairment in subacute stroke patients. Half of participants will see a video demonstrating the exercise to be performed before its actual execution, while the other half will see a video of a natural landscape followed by the same exercises the other group performs. All the patients will receive additional usual treatment.

DETAILED DESCRIPTION:
In this study, the intervention will be conducted using a system composed by multiple devices, which are:

* HTC Vive (HTC, headset e Steam station): three-dimensional viewer used for the implementation of the immersive virtual environment, allows both the visualization of the videos and of the exercises to be performed;
* Leap Motion Controller (infrared camera): contactless device for tracking the movement of the patient's fingers and hand;
* Zed Mini (RGB binocular camera and depth camera): Stereo Labs' Zed Mini stereoscopic camera is mounted on the HTC Vive viewer to allow virtual elements to be overlapped within the environment;
* Cometa Wavetrack (transmitter/receiver and Inertial Measurement Units): system for upper limb movement tracking through the use of four wireless inertial sensors applied to the chest, to the arm and to the forearm of the participant through elastic bands and to the hand of the participant through skin-compatible double-sided adhesive patches.

All the devices have been tested to ensure safety of the participants and are provided with the appropriate documentation of declaration of conformity according to the European reference regulations. A careful risk analysis was carried out to ensure the safety of the participants.

All the devices will be working simultaneously during each session of treatment. For the experimental group, the instrumentation will be used to see the video of the exercises that the participants will be later asked to perform and to actually perform them; in the control group, it will be used to see a video of a natural landscape with a 180° perspective and to perform the same exercises than the experimental group.

The devices will be used both for the execution of the exercises both to collect information listed in the outcomes section as secondary outcomes: in particular, these information will be provided by the Leap Motion and by the Cometa Wavetrack devices.

ELIGIBILITY:
Inclusion Criteria:

* Participant who suffered from an ictus 3 to 6 months before (subacute phase);
* Baseline scoring of the Upper Extremity portion of the Fugl Meyer between 20 and 60.

Exclusion Criteria:

* Other neurological pathologies (including previous strokes);
* Visual field impairments;
* Neuropsychological deficits that prevents the understanding of the instructions or the execution of the treatment (e.g. aphasia, apraxia, neglect);
* Baseline scoring of the Mini Mental State Examination (MMSE) lower that 24 (MMSE < 24);
* Orthopaedic or musculoskeletal limitations that do not allow the execution of the treatment;
* Clinical instability;
* Inability to understand the instructions needed to perform the test and the planned evaluations;
* People with electronic medical devices such as pacemakers;
* Medical history of epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of Upper limb function | Baseline (T0) and at the end of the treatment (T1, after 4 weeks).
  Upper extremity portion of the Fugl Meyer (UE-FM). This scale measures the function of the upper limb in a range of 0 to 66 points. Higher values represent a better outcome.
Change of hand dexterity | Baseline (T0) and at the end of the treatment (T1, after 4 weeks).
  Box and Block test. This test examines hand dexterity measuring the number of wooden blocks the participant is able to move from one box to another with the paretic hand in 60 seconds. Higher values represent a better outcome.

SECONDARY OUTCOMES:
Change of autonomy | Baseline (T0) and at the end of the treatment (T1, after 4 weeks).
  Barthel Index. This scale measures the ability of the subject to perform activities of daily living. Range 0-100. Higher values represent a better outcome.
Change of quality of Life | Baseline (T0) and at the end of the treatment (T1, after 4 weeks).
  EuroQol-5D questionnaire. This questionnaire measures the quality of life. Range 5-15. Lower values represent a better outcome.
Change of level completed | Baseline (T0) and at the end of the treatment (T1, after 4 weeks).
  Most difficult level the participant is able to complete, from 1 to 6. Higher values represent a better performance.
Change of number of correct tasks | Baseline (T0) and at the end of the treatment (T1, after 4 weeks).
  Number of tasks the participants performs correctly. Higher values represent a better performance.
Change of reaction time | Baseline (T0) and at the end of the treatment (T1, after 4 weeks).
  Seconds from the appearance of the target to the start of the movement. Lower values represent a better outcome.
Change of interaction time | Baseline (T0) and at the end of the treatment (T1, after 4 weeks).
  Seconds from the appearance of the target to its reaching. Lower values represent a better outcome.
Change of mean time of exercise execution | Baseline (T0) and at the end of the treatment (T1, after 4 weeks).
  Seconds required for single exercise execution. Lower values represent a better outcome.
Level of Satisfaction | At the end of the treatment (4 weeks).
  Likert 1-5. This scale measures the level of satisfaction of the subject regarding the treatment. Higher values represent a better outcome.
Change of Hand Max Reaching Velocity | Baseline (T0) and at the end of the treatment (T1, after 4 weeks).
  Maximal velocity (meters/seconds) of the hand movement during reaching of the target. Higher values represent a better outcome.
Change of % Cycle Hand Max Velocity | Baseline (T0) and at the end of the treatment (T1, after 4 weeks).
  Dividing the interaction time between the hand and the object into 100 parts, it represents the moment in which the hand reaches the maximal velocity.
Change of Mean SPARC | Baseline (T0) and at the end of the treatment (T1, after 4 weeks).
  Spectral parameter related to the smoothness of the movement. Negative values lower than -1 stand for lower smoothness.
Change of Mean Reach Path Ratio | Baseline (T0) and at the end of the treatment (T1, after 4 weeks).
  Parameter calculated as total distance traveled by the wrist of the subject divided by the length of a straight-line path from the reach's starting point (hand resting on the table) to ending point (target). Values equal or close to +1 represent a straight trajectory, while higher values stand for a more curved one.
Change of Tip Max Distance | Baseline (T0) and at the end of the treatment (T1, after 4 weeks).
  Maximal distance between the thumb and index fingertips.
Change of Tip Max Velocity | Baseline (T0) and at the end of the treatment (T1, after 4 weeks).
  Maximal velocity of opening and closing between the thumb and index fingertips.

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Buraschi, DPT, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi
Locations (1):
- Fondazione Don Carlo Gnocchi Onlus - Centro Ettore Spalenza, Rovato, Brescia, Italy

REFERENCES:
- [Background] Pollock A, Farmer SE, Brady MC, Langhorne P, Mead GE, Mehrholz J, van Wijck F. Interventions for improving upper limb function after stroke. Cochrane Database Syst Rev. 2014 Nov 12;2014(11):CD010820. doi: 10.1002/14651858.CD010820.pub2. PMID 25387001
- [Background] Laver KE, Lange B, George S, Deutsch JE, Saposnik G, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2017 Nov 20;11(11):CD008349. doi: 10.1002/14651858.CD008349.pub4. PMID 29156493
- [Background] Borges LR, Fernandes AB, Melo LP, Guerra RO, Campos TF. Action observation for upper limb rehabilitation after stroke. Cochrane Database Syst Rev. 2018 Oct 31;10(10):CD011887. doi: 10.1002/14651858.CD011887.pub2. PMID 30380586
- [Background] Shih TY, Wu CY, Lin KC, Cheng CH, Hsieh YW, Chen CL, Lai CJ, Chen CC. Effects of action observation therapy and mirror therapy after stroke on rehabilitation outcomes and neural mechanisms by MEG: study protocol for a randomized controlled trial. Trials. 2017 Oct 4;18(1):459. doi: 10.1186/s13063-017-2205-z. PMID 28978349
- [Background] Kim C-H, Bang D-H. Action observation training enhances upper extremity function in subacute stroke survivor with moderate impairment: a double-blind, randomized controlled pilot trial. J Korean Soc Phys Med. 2016;11(1):133-140. doi:10.13066/kspm.2016.11.1.133
- [Background] Franceschini M, Ceravolo MG, Agosti M, Cavallini P, Bonassi S, Dall'Armi V, Massucci M, Schifini F, Sale P. Clinical relevance of action observation in upper-limb stroke rehabilitation: a possible role in recovery of functional dexterity. A randomized clinical trial. Neurorehabil Neural Repair. 2012 Jun;26(5):456-62. doi: 10.1177/1545968311427406. Epub 2012 Jan 10. PMID 22235059
- [Background] Lin KC, Chuang LL, Wu CY, Hsieh YW, Chang WY. Responsiveness and validity of three dexterous function measures in stroke rehabilitation. J Rehabil Res Dev. 2010;47(6):563-71. doi: 10.1682/jrrd.2009.09.0155. PMID 20848369
- [Background] Kuk EJ, Kim JM, Oh DW, Hwang HJ. Effects of action observation therapy on hand dexterity and EEG-based cortical activation patterns in patients with post-stroke hemiparesis. Top Stroke Rehabil. 2016 Oct;23(5):318-25. doi: 10.1080/10749357.2016.1157972. Epub 2016 Mar 31. PMID 27077994
- [Background] Desrosiers J, Bravo G, Hebert R, Dutil E, Mercier L. Validation of the Box and Block Test as a measure of dexterity of elderly people: reliability, validity, and norms studies. Arch Phys Med Rehabil. 1994 Jul;75(7):751-5. PMID 8024419
- [Background] Fu J, Zeng M, Shen F, Cui Y, Zhu M, Gu X, Sun Y. Effects of action observation therapy on upper extremity function, daily activities and motion evoked potential in cerebral infarction patients. Medicine (Baltimore). 2017 Oct;96(42):e8080. doi: 10.1097/MD.0000000000008080. PMID 29049194
- [Background] Saposnik G, Cohen LG, Mamdani M, Pooyania S, Ploughman M, Cheung D, Shaw J, Hall J, Nord P, Dukelow S, Nilanont Y, De Los Rios F, Olmos L, Levin M, Teasell R, Cohen A, Thorpe K, Laupacis A, Bayley M; Stroke Outcomes Research Canada. Efficacy and safety of non-immersive virtual reality exercising in stroke rehabilitation (EVREST): a randomised, multicentre, single-blind, controlled trial. Lancet Neurol. 2016 Sep;15(10):1019-27. doi: 10.1016/S1474-4422(16)30121-1. Epub 2016 Jun 27. PMID 27365261
- [Background] Dorman PJ, Waddell F, Slattery J, Dennis M, Sandercock P. Is the EuroQol a valid measure of health-related quality of life after stroke? Stroke. 1997 Oct;28(10):1876-82. doi: 10.1161/01.str.28.10.1876. PMID 9341688
- [Background] Franceschini M, La Porta F, Agosti M, Massucci M; ICR2 group. Is health-related-quality of life of stroke patients influenced by neurological impairments at one year after stroke? Eur J Phys Rehabil Med. 2010 Sep;46(3):389-99. Epub 2010 Apr 13. PMID 20927005
- [Background] Lee KW, Kim SB, Lee JH, Lee SJ, Kim JW. Effect of Robot-Assisted Game Training on Upper Extremity Function in Stroke Patients. Ann Rehabil Med. 2017 Aug;41(4):539-546. doi: 10.5535/arm.2017.41.4.539. Epub 2017 Aug 31. PMID 28971037
- [Background] Langhorne P, Coupar F, Pollock A. Motor recovery after stroke: a systematic review. Lancet Neurol. 2009 Aug;8(8):741-54. doi: 10.1016/S1474-4422(09)70150-4. PMID 19608100